CLINICAL TRIAL: NCT07384949
Title: Correlation of Invasion Depth and Histopathological Features With Dermoscopic Findings in Cutaneous Squamous Cell Carcinoma
Brief Title: Correlation of Dermoscopic Findings With Histopathological Features and Invasion Depth in Cutaneous Squamous Cell Carcinoma
Acronym: SCC-DERM
Status: Not yet recruiting | Type: Observational
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Selma Nur Sahin, Dermatology Resident, MD, Istanbul Training and Research Hospital
Other Study IDs: ISTEAH-SCC-DERM-01
Record Dates: First submitted 2026-01-27; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Cutaneous Squamous Cell Cancer
Keywords: dermoscopy; Dermoscopic features; Histopathology correlation; Tumor invasion depth; Skin cancer imaging; Computer-assisted image analysis; Squamous cell carcinoma
MeSH Terms: conditions — Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cutaneous Squamous Cell Carcinoma Patients: This cohort includes patients diagnosed with cutaneous squamous cell carcinoma between 2016 and 2025 who underwent total excision and had available clinical, dermoscopic, and histopathological data in hospital records. No additional interventions were performed as part of the study.

SUMMARY:
This is a retrospective study including patients diagnosed with cutaneous squamous cell carcinoma between 2016 and 2025. Demographic, clinical, histopathological, and dermoscopic data were obtained from hospital records. Dermoscopic images taken with the FotoFinder dermoscope were independently evaluated by two dermatologists in a blinded manner. In addition, images were labeled using computer software and analyzed to measure the proportion of specific dermoscopic structures within the total lesion area. These quantitative data were used to examine the relationship between dermoscopic features and histopathological findings.

DETAILED DESCRIPTION:
This retrospective study includes patients who were diagnosed with cutaneous squamous cell carcinoma (cSCC) and underwent total excision between 2016 and 2025 at a tertiary dermatology center. Patient data were obtained from the hospital electronic medical record system, including demographic characteristics (age, sex), clinical features (lesion location, size, and morphology), and histopathological parameters such as tumor depth of invasion and histopathological subtype.

Dermoscopic images were acquired using a FotoFinder digital dermoscope as part of routine clinical documentation prior to excision. All dermoscopic images were independently evaluated by two dermatologists who were blinded to the histopathological results. Dermoscopic features, including vascular patterns and keratin-related structures, were recorded according to predefined criteria. Interobserver agreement was assessed, and discordant evaluations were resolved by consensus.

For objective image analysis, dermoscopic images were segmented and annotated using the LabelMe software. Regions of interest corresponding to specific dermoscopic structures were manually labeled, and pixel-based quantitative measurements were extracted using computer-assisted image analysis pipelines developed in the Visual Studio Code environment. The proportional area of each dermoscopic structure relative to the total lesion surface was calculated and recorded as numerical data.

The primary objective of the study is to investigate the relationship between dermoscopic features and histopathological parameters, particularly tumor invasion depth and histopathological subtype. Secondary objectives include assessing whether quantitative dermoscopic measurements can improve the prediction of invasive behavior in cSCC.

Statistical analyses will be performed to evaluate correlations between dermoscopic variables and histopathological outcomes. Appropriate parametric or non-parametric tests will be used depending on data distribution. Multivariate analyses may be conducted to identify independent dermoscopic predictors of deeper tumor invasion. All analyses will be performed using standard statistical software.

As this is a retrospective study using existing clinical data and images, no additional interventions or patient contact are involved. All data will be anonymized prior to analysis in accordance with institutional and ethical regulations.

ELIGIBILITY:
Inclusion Criteria:Age between 18 and 100 years at the time of diagnosis

Histopathologically confirmed cutaneous squamous cell carcinoma

Lesions that underwent total surgical excision

Histopathology reports including both tumor differentiation grade and invasion depth

Availability of dermoscopic images obtained prior to excision

Dermoscopic images of sufficient quality for evaluation and image analysis -

Exclusion Criteria:

Lesions that received any prior treatment, including radiotherapy, chemotherapy, cryotherapy, or other destructive or topical treatments before excision

Incomplete clinical, dermoscopic, or histopathological data

Poor-quality dermoscopic images not suitable for reliable evaluation or segmentation

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 to 100 years who were diagnosed with cutaneous squamous cell carcinoma and treated with total surgical excision between 2016 and 2025. Only cases with complete clinical, dermoscopic, and histopathological records, including documented tumor differentiation and invasion depth, were included. No additional diagnostic or therapeutic procedures were performed as part of the study.
Sampling Method: Non-Probability Sample
Enrollment: 238 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Correlation between dermoscopic features and tumor invasion depth | Retrospective analysis of records from 2016 to 2025
  The association between predefined dermoscopic features and histopathological tumor invasion depth will be evaluated using quantitative and qualitative dermoscopic assessments.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Istanbul Training and Research Hospital, Department of Dermatology, Istanbul, FATİH, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to patient confidentiality, institutional data protection policies, and the retrospective nature of the study. All analyses will be reported in aggregate form only.